CLINICAL TRIAL: NCT03331731
Title: A Multi-centre Phase II Study to Determine the Response Kinetics, Safety and Efficacy of Pembrolizumab as Frontline Treatment of Patients With Hodgkin Lymphoma Considered Unsuitable for ABVD
Brief Title: A Phase II Study to Determine Pembrolizumab as Frontline Treatment of Patients With Hodgkin Lymphoma
Acronym: PLIMATH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/158
Record Dates: First submitted 2017-10-10; First posted 2017-11-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single arm, open label, phase II, international, multicentre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single Arm
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to test how safe and effective the research study drug, pembrolizumab is as a treatment for patients with Hodgkin lymphoma who have not previously been treated for this disease and are unsuitable for standard treatment (adriamycin, bleomycin, vinblastine, dacarbazine ABVD).

DETAILED DESCRIPTION:
The study is a single arm, open label, phase II, international, multi-centre study. Sample size will be 25 evaluable patients with a recruitment period of 2 years. Patients will be administered 200mg pembrolizumab IV every 3 weeks up to 35 cycles or 2 years. Patients will be followed-up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent for the trial.
2. Be 18 years or greater on day of signing informed consent.
3. Have a diagnosis of Hodgkin lymphoma.
4. The patient must meet one of the following criteria:

   1. Age ≥65
   2. Considered by the investigator to be ineligible for front-line ABVD combination chemotherapy due to reasons of medical co-morbidity
5. Have measurable disease based on the Lugano classification
6. Have stage III or IV disease; or disease stage II disease that cannot be irradiated without unacceptable toxicity in the view of the investigator and patient.
7. Be willing to provide tissue from a "newly-obtained" core or excisional biopsy of a tumour lesion. Newly-obtained is defined as a specimen obtained up to 8 weeks (56 days) prior to registration. Patients for whom newly-obtained samples cannot be provided (e.g. inaccessible or patient safety concern) may submit an archived specimen only upon agreement from the CPI.
8. Have a performance status of 0, 1 or 2 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined in Table 2, all screening labs should be performed within 10 days of registration.
10. Female patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female patients of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 7.14 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
12. Male patients of childbearing potential must agree to use an adequate method of contraception as outlined in Section 7.14 - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of registration.
2. Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days of registration. Is taking chronic systemic steroids (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to registration.

   Note: Apart from steroids for palliative purposes specifically for lymphoma-associated symptoms (prednisolone 50mg or equivalent for up to 10 doses) or patients with asthma or chronic obstructive pulmonary disease that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (MoAb) within 4 weeks prior to registration or who has not recovered (i.e., ≤ Grade 1 at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If a patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to registration.
7. Subject has a history of other active malignancies other than HL within the past 2 years prior to study entry, with the exception of:

   * Adequately treated carcinoma in situ of the cervix uteri
   * Adequately treated basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically resected (or treated with other modalities) with curative intent and less than 10% risk of recurrence in next 12 months.
   * Untreated monoclonal B lymphocytosis or chronic lymphocytic leukaemia stage 0 with <50% increase in lymphocyte count in preceding 6 months or absolute lymphocyte count of <10 x10^9/L.
   * Myelodysplastic syndrome with no excess of blasts and blood count parameters meeting inclusion criteria, with no prior disease-modifying therapy.
   * Low-risk early stage prostate adenocarcinoma (T1-T2aN0M0 and Gleason score ≤6 and PSA ≤10ng/mL) for which the management plan is active surveillance, or prostate adenocarcinoma with biochemical-only recurrence with documented PSA doubling time of > 12 months for which the management plan is active surveillance
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has a history of non-infectious pneumonitis that required steroids or has current pneumonitis.
10. Has an active infection requiring systemic therapy more than oral antibiotics.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent in the preceding 12 months.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days of registration. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
18. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to registration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to registration. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Response using Lugano Criteria | At each treatment cycle 1 to 35 (each cycle is 3 weeks)
  Response will be assessed by Lugano criteria. Overall response is defined as achieving either CR or PR at any stage from time of commencement of protocol treatment to time of treatment cessation for whatever reason.

SECONDARY OUTCOMES:
Response using LYRIC Criteria | At each treatment cycle 1 to 35 (each cycle is 3 weeks)
  Response will be assessed by LYRIC criteria
Adverse Events | Screening, Cycles 1-35 (each cycle is 3 weeks), end of treatment (2 years), 30 days from date of last dose, up until the first sign of progression through to study completion (3 years)
  Adverse Events will be evaluated using CTCAE version 4.03 as worst grade per AE
Progression Free Survival (PFS) | up until the first sign of progression through to study completion (3 years)
  PFS will be measured from the date of treatment commencement to the date of first progression at any site or date of death from any cause
Overal Survival (OS) | up until the first sign of progression through to study completion (3 years)
  OS will be measured from the date of treatment commencement to the date death from any cause.
Treatment Intensity | At each treatment cycle 1 to 35 (each cycle is 3 weeks)
  Treatment intensity will be defined as the actual total dose received divided by the actual treatment period
Event Free Survival (EFS) | up until the first sign of progression through to study completion (3 years)
  EFS will be measured from the date of treatment commencement to date of documented disease progression at any site, date of commencement of next-line treatment, or date of death from any cause, whichever occurs first.
Duration of response (DoR) | up until the first sign of progression through to study completion (3 years)
  DoR will be assessed on patients who responded to treatment and will be measured from the date of first documented disease response to the earliest recurrence or progressive disease. Deceased patients without recurrence or progressive disease will be censored at the last disease assessment date.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (6):
- Australia (5):
  - Concord Hospital, Concord, New South Wales
  - Linear Clinical Research, Nedlands, Perth
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No